CLINICAL TRIAL: NCT04203095
Title: Dynamic Monitor of Serum Chromosomal Instability Detected by UCAD as a Surrogate Biomarker of Treatment Efficacy in PD1 Inhibitor Based Immunotherapy for Lung Cancer Patients
Brief Title: Chromosomal Instability as a Surrogate Biomarker of Drug Resistance in Immunotherapy for Lung Cancer Patients
Acronym: CINSBDRILCP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Di Zheng, Director of medical oncology, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: ph-pg001
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Lung Cancer
Keywords: Chromosomal aneuploidy detection; lung cancer; PD-1/PD-L1; Drug resistance in Immunotherapy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The extracted cell free DNA from peripheral blood will be analyzed by Ultrasensitive Chromosomal Aneuploidy Detection to determine the level of chromosomal instability.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient with PD1 antibody treatment: Investigators will detect cfDNA CIN of lung cancer patients 1day (Day 0) before treatment with PD1 antibody, then Day 22 and Day 64 after treatment with PD1 antibody, as well as at the time of disease progression confirmed.
  The correlation of CIN and drug resistance to PD1 antibody was analyzed.
  Interventions: Diagnostic Test: the level of plasma cfDNA CINs

INTERVENTIONS:
Diagnostic Test: the level of plasma cfDNA CINs — The extracted cfDNA from PB will be analyzed by UCAD to determine the level of CINs.

SUMMARY:
PD1, as an immune checkpoint inhibitor, has provided a new therapeutic approach for patients with cancer, including patients. Although immunotherapy has proven effective, most patients do not benefit from it because of a large proportion which developing primary and acquired resistance. However, there is still a lack of accurate and effective molecular biomarkers to accurately evaluate the drug resistance of patients treated with immune checkpoint inhibitors (ICI), so as to maximize the therapeutic effect in patients. Chromosomal instability (CIN) is one of the most prominent and common characteristics of solid tumors, accelerating the development of anti-cancer drug resistance, often leading to treatment failure and disease recurrence, which limits the effectiveness of most current treatments. Hence the aim of this study is to evaluate dynamic CIN continuously monitored in the blood of patients with lung cancer treated with ICIs with Ultrasensitive Chromosomal Aneuploidy Detection (UCAD) to establish a new molecular immune resistance evaluation index. Further, the correlation between the evolution of tumor cloning and ICI resistance in patients during treatment was analyzed based on the results of dynamic CIN detection. This not only evaluate the efficacy of the ICI treatment in real-time, but also enables better understanding and overcoming the resistance mechanism of immunotherapy in the future.

DETAILED DESCRIPTION:
Immune checkpoint inhibitors (ICI) targeted to PD-1/PD-L1 axis has a higher response rate and lower incidence of side effects compared with anti-CTLA4, and has been proved to have survival advantages in many different malignant tumors, which has been approved as a second-line or first-line treatment for a growing number of malignancies, including lung cancer. As results of retrospective analysis led by Roberto Ferrara, although the efficacy of ICI treatment is obvious in non-small cell lung cancer (NSCLC), there are significant differences in efficacy and responsiveness in different patients. Therefore, establishing predictive biomarkers for immunotherapy is the key to maximizing the therapeutic effect and studying drug resistance. According to clinical trial data after immunotherapy, there are three main groups: (1) those who respond initially and continue to respond (responders); (2) those who have never responded (primary resistance); (3) Those who initially respond but eventually develop into disease progression (secondary resistance).Currently, PD-L1 expression is one of the most common biomarkers for immunotherapy, PD-L1 expression itself does not accurately predict immunotherapy response, due to that the many patients with higher PD-L1 have no response to clinical treatment, and many patients with lower PD-L1 respond better. Although tumor mutation burden (TMB ) used as a biomarker for the treatment of NSCLC by Opdivo could better differentiate the people who benefit compared with PD-L1, however, TMB as a biomarker to determine the criteria for the application of ICI treatment resistance is also limited because of its specific mechanism involved in tumor immune regulation needs to be further clarified and high cost of TMB detection using NGS for whole exome sequencing analysis.

As one of the most prominent and common features of solid tumors, chromosomal instability (CIN) accelerates the development of anticancer drug resistance, often leading to treatment failure and disease recurrence, which limits the effectiveness of most current treatments. Previous studies have shown that CIN promotes the emergence of multidrug resistance by providing higher levels of genetic diversity, leading to multidrug resistance. In NSCLC, the researchers found that genomic doubling and sustained dynamic CIN were associated with intratumoral heterogeneity and led to parallel evolution of CDNAs, including CDK4, FOXA1, and BCL11A. It is worth noting that the study found consistency in the variation of mutation levels, indicating that CIN in lung cancer is more likely to select driving events than other mutation processes. CIN enables cells to enter several different evolutionary trajectories and adapt to the selective pressure generated by treatment, which is the basis of drug resistance. Based on the above, CIN may become a more accurate and effective biomarker for the study of drug resistance mechanism of ICI in lung cancer. NGS technology can obtain more comprehensive genomic information while detecting cost reduction, making CIN detection more accurate and practical than FISH used for evaluating CIN in patient commonly.As a new Detection method based on NGS technology, Ultrasensitive Chromosomal Aneuploidy Detection (UCAD) has been developed in our previous study. In which, low-coverage whole-genome sequencing technology based on NGS was adopted to detect CIN of ctDNA in patients' peripheral blood, and bioinformatics analysis was performed to determine the risk of malignancy (or recurrence) and the extent of tumor burden and CIN. It has important clinical value in auxiliary diagnosis, therapeutic effect monitoring, recurrence and metastasis monitoring and prognosis evaluation of tumor patients.

This study proposes that continuous dynamic CIN is related to intratumor heterogeneity, which drives parallel evolution of somatic copy-number alterations (SCNAs) and promotes the emergence of drug-resistant clones by providing a higher level of genetic diversity of tumor cells, thus leading to drug resistance in patients treated with ICI. Investigators aimed to continuously monitor dynamic CIN in the blood of patients with lung cancer after second-line treatment with UCAD to establish a new molecular immune resistance evaluation index. Further, the correlation between the evolution of tumor cloning and ICI resistance in patients during treatment was analyzed based on the detection results of dynamic CIN.

ELIGIBILITY:
Inclusion Criteria:

* Stage IIIa-IVb Non-small-cell lung cancer patients without EGFR，ALK,ROS1,c-Met driven gene mutation. Male or female patients aged 20-70 years.
* Patients planed to receive PD1 antibody treatment with or without chemotherapy, including as the neo-adjuvant therapy.
* The subjects' age, sex, marital and reproductive history, collection time, pathology, cytology and imaging diagnosis were complete.
* Participants signed informed consent form.

Exclusion Criteria:

* Eligible to target therapy with driven gene mutation.
* Without measurable target lesion according to the RECIST criteria.
* Age under 20 years or more than 70.
* Individuals unwilling to sign the consent form or unwilling to provide PB for test or unwilling to provide the medical record.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with lung cancer in Shanghai Pulmonary Hospital (SPH) from Aug 2019 till the end of this study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-11-10 (Actual); Primary Completion 2020-11-11 (Estimated); Study Completion 2021-11-11 (Estimated)

PRIMARY OUTCOMES:
the concordance bettwen CINs and treatment outcomes The concordance between CINs and treatment outcomes | through study completion, an average of 3 months
  According to the correlation analysis between the patient's clinical drug resistance and CIN detected using UCAD, the stratified cutoff value interval of the patient was found, which was divided into four treatment outcomes based on CIN assessment : significant efficacy, primary drug resistance, acquired drug resistance and possible super progress.

SECONDARY OUTCOMES:
the concordance bettwen CINs and clinical monitoring | through study completion, an average of 3 months
  Analyze the correlation between the dynamic change of CIN using UCAD and the efficacy evaluation by the RECIST criteria , and compare the time difference and accuracy between UCAD and imaging test and serology.

CONTACTS AND LOCATIONS:
Overall Officials: Di Zheng, PhD, Study Director — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Di Zheng, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pardoll DM. The blockade of immune checkpoints in cancer immunotherapy. Nat Rev Cancer. 2012 Mar 22;12(4):252-64. doi: 10.1038/nrc3239. PMID 22437870
- [Background] Brahmer JR, Tykodi SS, Chow LQ, Hwu WJ, Topalian SL, Hwu P, Drake CG, Camacho LH, Kauh J, Odunsi K, Pitot HC, Hamid O, Bhatia S, Martins R, Eaton K, Chen S, Salay TM, Alaparthy S, Grosso JF, Korman AJ, Parker SM, Agrawal S, Goldberg SM, Pardoll DM, Gupta A, Wigginton JM. Safety and activity of anti-PD-L1 antibody in patients with advanced cancer. N Engl J Med. 2012 Jun 28;366(26):2455-65. doi: 10.1056/NEJMoa1200694. Epub 2012 Jun 2. PMID 22658128
- [Background] Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, Powderly JD, Carvajal RD, Sosman JA, Atkins MB, Leming PD, Spigel DR, Antonia SJ, Horn L, Drake CG, Pardoll DM, Chen L, Sharfman WH, Anders RA, Taube JM, McMiller TL, Xu H, Korman AJ, Jure-Kunkel M, Agrawal S, McDonald D, Kollia GD, Gupta A, Wigginton JM, Sznol M. Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med. 2012 Jun 28;366(26):2443-54. doi: 10.1056/NEJMoa1200690. Epub 2012 Jun 2. PMID 22658127
- [Background] Wan MT, Ming ME. Nivolumab versus ipilimumab in the treatment of advanced melanoma: a critical appraisal: ORIGINAL ARTICLE: Wolchok JD, Chiarion-Sileni V, Gonzalez R et al. Overall survival with combined nivolumab and ipilimumab in advanced melanoma. N Engl J Med 2017; 377:1345-56. Br J Dermatol. 2018 Aug;179(2):296-300. doi: 10.1111/bjd.16785. Epub 2018 Jun 5. PMID 29766492
- [Background] Sharma P, Hu-Lieskovan S, Wargo JA, Ribas A. Primary, Adaptive, and Acquired Resistance to Cancer Immunotherapy. Cell. 2017 Feb 9;168(4):707-723. doi: 10.1016/j.cell.2017.01.017. PMID 28187290
- [Background] Gong J, Chehrazi-Raffle A, Reddi S, Salgia R. Development of PD-1 and PD-L1 inhibitors as a form of cancer immunotherapy: a comprehensive review of registration trials and future considerations. J Immunother Cancer. 2018 Jan 23;6(1):8. doi: 10.1186/s40425-018-0316-z. PMID 29357948
- [Background] Estin CD, Stevenson U, Kahn M, Hellstrom I, Hellstrom KE. Transfected mouse melanoma lines that express various levels of human melanoma-associated antigen p97. J Natl Cancer Inst. 1989 Mar 15;81(6):445-8. doi: 10.1093/jnci/81.6.445. PMID 2918553
- [Background] Restifo NP, Smyth MJ, Snyder A. Acquired resistance to immunotherapy and future challenges. Nat Rev Cancer. 2016 Feb;16(2):121-6. doi: 10.1038/nrc.2016.2. PMID 26822578
- [Background] O'Donnell JS, Long GV, Scolyer RA, Teng MW, Smyth MJ. Resistance to PD1/PDL1 checkpoint inhibition. Cancer Treat Rev. 2017 Jan;52:71-81. doi: 10.1016/j.ctrv.2016.11.007. Epub 2016 Nov 27. PMID 27951441
- [Background] Haratani K, Hayashi H, Tanaka T, Kaneda H, Togashi Y, Sakai K, Hayashi K, Tomida S, Chiba Y, Yonesaka K, Nonagase Y, Takahama T, Tanizaki J, Tanaka K, Yoshida T, Tanimura K, Takeda M, Yoshioka H, Ishida T, Mitsudomi T, Nishio K, Nakagawa K. Tumor immune microenvironment and nivolumab efficacy in EGFR mutation-positive non-small-cell lung cancer based on T790M status after disease progression during EGFR-TKI treatment. Ann Oncol. 2017 Jul 1;28(7):1532-1539. doi: 10.1093/annonc/mdx183. PMID 28407039
- [Background] Sansregret L, Vanhaesebroeck B, Swanton C. Determinants and clinical implications of chromosomal instability in cancer. Nat Rev Clin Oncol. 2018 Mar;15(3):139-150. doi: 10.1038/nrclinonc.2017.198. Epub 2018 Jan 3. PMID 29297505
- [Background] Lee AJ, Endesfelder D, Rowan AJ, Walther A, Birkbak NJ, Futreal PA, Downward J, Szallasi Z, Tomlinson IP, Howell M, Kschischo M, Swanton C. Chromosomal instability confers intrinsic multidrug resistance. Cancer Res. 2011 Mar 1;71(5):1858-70. doi: 10.1158/0008-5472.CAN-10-3604. PMID 21363922
- [Background] Kuznetsova AY, Seget K, Moeller GK, de Pagter MS, de Roos JA, Durrbaum M, Kuffer C, Muller S, Zaman GJ, Kloosterman WP, Storchova Z. Chromosomal instability, tolerance of mitotic errors and multidrug resistance are promoted by tetraploidization in human cells. Cell Cycle. 2015;14(17):2810-20. doi: 10.1080/15384101.2015.1068482. PMID 26151317
- [Background] Jamal-Hanjani M, Wilson GA, McGranahan N, Birkbak NJ, Watkins TBK, Veeriah S, Shafi S, Johnson DH, Mitter R, Rosenthal R, Salm M, Horswell S, Escudero M, Matthews N, Rowan A, Chambers T, Moore DA, Turajlic S, Xu H, Lee SM, Forster MD, Ahmad T, Hiley CT, Abbosh C, Falzon M, Borg E, Marafioti T, Lawrence D, Hayward M, Kolvekar S, Panagiotopoulos N, Janes SM, Thakrar R, Ahmed A, Blackhall F, Summers Y, Shah R, Joseph L, Quinn AM, Crosbie PA, Naidu B, Middleton G, Langman G, Trotter S, Nicolson M, Remmen H, Kerr K, Chetty M, Gomersall L, Fennell DA, Nakas A, Rathinam S, Anand G, Khan S, Russell P, Ezhil V, Ismail B, Irvin-Sellers M, Prakash V, Lester JF, Kornaszewska M, Attanoos R, Adams H, Davies H, Dentro S, Taniere P, O'Sullivan B, Lowe HL, Hartley JA, Iles N, Bell H, Ngai Y, Shaw JA, Herrero J, Szallasi Z, Schwarz RF, Stewart A, Quezada SA, Le Quesne J, Van Loo P, Dive C, Hackshaw A, Swanton C; TRACERx Consortium. Tracking the Evolution of Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Jun 1;376(22):2109-2121. doi: 10.1056/NEJMoa1616288. Epub 2017 Apr 26. PMID 28445112
- [Background] Xue Y, Martelotto L, Baslan T, Vides A, Solomon M, Mai TT, Chaudhary N, Riely GJ, Li BT, Scott K, Cechhi F, Stierner U, Chadalavada K, de Stanchina E, Schwartz S, Hembrough T, Nanjangud G, Berger MF, Nilsson J, Lowe SW, Reis-Filho JS, Rosen N, Lito P. An approach to suppress the evolution of resistance in BRAFV600E-mutant cancer. Nat Med. 2017 Aug;23(8):929-937. doi: 10.1038/nm.4369. Epub 2017 Jul 17. PMID 28714990
- [Background] Juric D, Castel P, Griffith M, Griffith OL, Won HH, Ellis H, Ebbesen SH, Ainscough BJ, Ramu A, Iyer G, Shah RH, Huynh T, Mino-Kenudson M, Sgroi D, Isakoff S, Thabet A, Elamine L, Solit DB, Lowe SW, Quadt C, Peters M, Derti A, Schegel R, Huang A, Mardis ER, Berger MF, Baselga J, Scaltriti M. Convergent loss of PTEN leads to clinical resistance to a PI(3)Kalpha inhibitor. Nature. 2015 Feb 12;518(7538):240-4. doi: 10.1038/nature13948. Epub 2014 Nov 17. PMID 25409150
- [Background] Heng HH, Spyropoulos B, Moens PB. FISH technology in chromosome and genome research. Bioessays. 1997 Jan;19(1):75-84. doi: 10.1002/bies.950190112. PMID 9008419